CLINICAL TRIAL: NCT00847782
Title: An Experimental Medicine Study to Quantify PCSK9 Serum Concentrations and LDL Receptor Expression in Peripheral Blood Cells in Normal and Hypercholesterolemic Subjects
Brief Title: An Experimental Medicine Study to Evaluate Serum Biomarkers of Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CV198-001
Record Dates: First submitted 2009-02-06; First posted 2009-02-19 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blood draw (Group 1) (Other): Normocholesterolemic Subjects
  Normal Healthy Volunteers
  Interventions: Procedure: Blood draw
- Blood draw (Group 2) (Other): Hypercholesterolemic Subjects
  Interventions: Procedure: Blood draw
- Blood draw (Group 3) (Other): Hypercholesterolemic Subjects with Statin Treatment
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — 1 day

SUMMARY:
The purpose of this study is to validate novel assays for serum biomarkers of lipid metabolism (PCSK9 and LDL receptor) and to obtain information about how these biomarkers differ in subjects with normal or high cholesterol levels

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia
* Statin monotherapy

Exclusion Criteria:

* Significant acute or chronic illness
* Secondary causes of hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Serum PCSK9 concentration | Initial assessment will occur when Group 1 has 50 subjects enrolled and Groups 2 and 3 have 30 subjects enrolled

SECONDARY OUTCOMES:
Serum LDL cholesterol concentration | Initial assessment will occur when Groups 2 and 3 have enrolled 30 subjects
Serum HDL cholesterol concentration | Initial assessment will occur when Groups 2 and 3 have enrolled 30 subjects
Serum TG concentration | Initial assessment will occur when Groups 2 and 3 have enrolled 30 subjects
Serum Apo B concentration | Initial assessment will occur when Groups 2 and 3 have enrolled 30 subjects

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Montreal, Quebec, Canada

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx